CLINICAL TRIAL: NCT00486434
Title: A Randomized, Double-Blind, Multi-Center, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Salmon Calcitonin in the Treatment of Subjects With Knee Osteoarthritis
Brief Title: Efficacy and Safety of Oral Salmon Calcitonin in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Bioscience A/S (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSMC021C2301
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, oral salmon calcitonin, treatment, efficacy, tolerability
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): SMC021 Oral Calcitonin, 0.8 mg twice daily during 24 months
  Interventions: Drug: SMC021 Oral Calcitonin
- 2 (Placebo Comparator): SMC021 Placebo, orally twice daily during 24 months
  Interventions: Drug: SMC021 Placebo

INTERVENTIONS:
Drug: SMC021 Oral Calcitonin — 0.8mg SMC021 (Oral Calcitoinin) twice daily
  Arms: 1
Drug: SMC021 Placebo — Placebo orally, twice daily
  Arms: 2

SUMMARY:
The purpose of this Phase III study is to evaluate the efficacy and safety of oral salmon calcitonin in the treatment of patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Medical history and symptoms of knee osteoarthritis

Exclusion Criteria:

* Any other disease or medication affecting the bone or cartilage.
* Any clinical signs or laboratory evidence diseases, which in the Investigator's opinion would preclude the participant from adhering to the Protocol or completing the trial.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 51 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1176 (Actual)
Dates: Start 2007-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bente J Riis, M.D., Study Chair — Nordic Bioscience A/S
Locations (9):
- CCBR Czech, Pardubice, Czechia
- Denmark (3):
  - CCBR Aalborg, Aalborg
  - CCBR Ballerup, Ballerup Municipality
  - CCBR Vejle, Vejle
- CCBR Estonia, Tallinn, Estonia
- CCBR Hong Kong, Hong Kong, Hong Kong
- Poland (2):
  - Centrum Osteoporozy i Chorób Kostno Stawowych, ul. Waryńskiego 6/2, Bialystok
  - CCBR Poland, Warsaw
- CCBR Romania, Bucharest, Romania

REFERENCES:
- [Derived] Bihlet AR, Bjerre-Bastos JJ, Andersen JR, Byrjalsen I, Karsdal MA, Bay-Jensen AC. Clinical and biochemical factors associated with risk of total joint replacement and radiographic progression in osteoarthritis: Data from two phase III clinical trials. Semin Arthritis Rheum. 2020 Dec;50(6):1374-1381. doi: 10.1016/j.semarthrit.2020.03.002. Epub 2020 Mar 15. PMID 32249039
- [Derived] Bihlet AR, Byrjalsen I, Bay-Jensen AC, Andersen JR, Christiansen C, Riis BJ, Karsdal MA. Associations between biomarkers of bone and cartilage turnover, gender, pain categories and radiographic severity in knee osteoarthritis. Arthritis Res Ther. 2019 Sep 3;21(1):203. doi: 10.1186/s13075-019-1987-7. PMID 31481084
- [Derived] Bihlet AR, Byrjalsen I, Bay-Jensen AC, Andersen JR, Christiansen C, Riis BJ, Valter I, Karsdal MA, Hochberg MC. Identification of pain categories associated with change in pain in patients receiving placebo: data from two phase 3 randomized clinical trials in symptomatic knee osteoarthritis. BMC Musculoskelet Disord. 2018 Jan 17;19(1):17. doi: 10.1186/s12891-018-1938-5. PMID 29343266
- [Derived] Karsdal MA, Byrjalsen I, Alexandersen P, Bihlet A, Andersen JR, Riis BJ, Bay-Jensen AC, Christiansen C; CSMC021C2301/2 investigators. Treatment of symptomatic knee osteoarthritis with oral salmon calcitonin: results from two phase 3 trials. Osteoarthritis Cartilage. 2015 Apr;23(4):532-43. doi: 10.1016/j.joca.2014.12.019. Epub 2015 Jan 9. PMID 25582279
- [Derived] Henriksen K, Bay-Jensen AC, Christiansen C, Karsdal MA. Oral salmon calcitonin--pharmacology in osteoporosis. Expert Opin Biol Ther. 2010 Nov;10(11):1617-29. doi: 10.1517/14712598.2010.526104. Epub 2010 Oct 11. PMID 20932224

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Arm: 0.8mg SMC021 Oral Calcitonin tablet twice daily
- Placebo Arm: 1 SMC021 Placebo tablet twice daily
Period: Overall Study
Arm/Group | Active Arm | Placebo Arm
Started | 588 | 588
Completed | 394 | 454
Not Completed | 194 | 134
Not completed — Withdrawal by Subject | 34 | 39
Not completed — Adverse Event | 118 | 44
Not completed — Protocol Violation | 22 | 21
Not completed — Lack of Efficacy | 12 | 19
Not completed — Lost to Follow-up | 2 | 3
Not completed — Death | 1 | 2
Not completed — Personal reasons | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Placebo Arm | Total
Number analyzed (Participants) | 588 | 588 | 1176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 293 | 321 | 614
  >=65 years | 295 | 267 | 562
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (6.84) | 63.9 (6.41) | 64.0 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 418 | 386 | 804
  Male | 170 | 202 | 372
Region of Enrollment [Number; unit: participants]
  Hong Kong | 51 | 51 | 102
  Czech Republic | 47 | 48 | 95
  Estonia | 47 | 47 | 94
  Poland | 33 | 34 | 67
  Romania | 40 | 39 | 79
  Denmark | 370 | 369 | 739

OUTCOME MEASURES:

1. Primary Outcome: Joint Space Width (JSW) in the Medial Tibiofemoral Knee Joint in Signal Knee Measured by X-ray After 24 Months.
Description: The signal knee was chosen prior to randomization based on which knee met the inclusion and exclusion criteria. The JSW is the space measured in mm between the 2 bones in the knee joint and this is assessed by x-ray. The JSW decreases with disease progression. The lower limit for participation in the trial were 2 mm JSW. There were no upper limit as long as inclusion and exclusion criteria were met. The outcome was measured as a change in JSW from baseline to month 24.
Time Frame: Change from baseline to 24 months
Population: The number of participants analysed for this outcome is the intent-to-treat (ITT) population. ITT is the number of randomized subjects who received at least one dose of study medication. There were 7 patients in the randomized population who did not receive any study drug and where therefore excluded from the ITT analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 585 | 584
mm | -0.188 (0.5626) | -0.198 (0.5069)

2. Primary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Subscore in the Signal Knee
Description: WOMAC is a self-administered set of standardized questionnaires to evaluate the condition of patients with osteoarthritis of the knee. The subject marks on a scale (1-100) the pain associated with performing each daily activity listed in the questionnaire. 0 is no pain (best), 100 is extreme pain (Worst). The total function sub score for the questions are then calculated. Total possible minimum sub score is 0, maximum is 500. The final outcome is the absolute change from baseline to 24 months. If the outcome is less that 0 there is improvement (less pain).
Time Frame: Change from baseline to 24 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 585 | 584
Units on a scale | -124.0 [-391 to 218] | -109.0 [-410 to 349]

3. Primary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Function Subscore in the Signal Knee.
Description: WOMAC is a self-administered set of standardized questionnaires to evaluate the condition of patients with osteoarthritis of the knee. The subject marks on a scale (1-100) the degree of difficulty for performing each daily function listed in the questionnaire. 0 is no difficulty (best), 100 is extreme difficulty (worst). The total function sub score for the questions are then calculated. Total possible minimum sub score is 0, maximum is 1700. The final outcome is the absolute change from baseline to 24 months. If the outcome is less that 0 there is improvement (less difficulty).
Time Frame: Change from baseline to 24 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 585 | 584
Units on a scale | -390.0 [-1307 to 783] | -299.5 [-1342 to 915]

4. Secondary Outcome: Changes in Biochemical Markers of Bone & Cartilage Metabolism.
Description: The central laboratory analyzed serum CTX-I (S-Crosslaps, Elecsys) and osteocalcin as well as urine CTX-I/creatinine and CTX-II/creatinine. It was originally planned that serum CTX-II would be measured, but this was not done.
Time Frame: From Baseline to Month 24
Population: ITT Population. The number analyzed in some rows differs from the overall number analyzed due to missing values from patients who prematurely discontinued.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 585 | 584
percentage of change
  Serum CTX-I (ng/mL): number analyzed (Participants) | 578 | 577
  Serum CTX-I (ng/mL) | 41.358 (68.1153) | 62.883 (65.7225)
  Serum Osteocalcin (ng/mL): number analyzed (Participants) | 578 | 577
  Serum Osteocalcin (ng/mL) | -9.134 (22.1368) | 1.785 (22.8324)
  24-h urine CTX-I/creatinine (µg/mmol): number analyzed (Participants) | 574 | 571
  24-h urine CTX-I/creatinine (µg/mmol) | -8.959 (50.0723) | 8.311 (55.4934)
  24-h urine CTX-II/creatinine (ng/mmol): number analyzed (Participants) | 574 | 571
  24-h urine CTX-II/creatinine (ng/mmol) | 0.484 (56.4879) | 11.266 (49.6250)

5. Secondary Outcome: Effect on Hand Osteoarthritis (OA) Assessed by X-ray & Questionnaire From Baseline to 24 Months
Description: To assess disease progression of OA affected joints, X-rays of both hands were performed & assessed by two central readers (at Synarc). Hand OA was assessed by calculating total score for osteophytes, cyst erosion, & joint space narrowing, each of which were based on sum of left and right hand X-ray analysis with possible scores of 0-66. The overall total score (possible range 0-198) was also used. Higher scores (closer to 66 or to 198 when using overall total score) imply a worse outcome. Hand analyses were based on double readings, and the mean was used in the analyses.
  The AUStralian/CANadian Osteoarthritis Hand Index (AUSCAN) questionnaire was also used for assessment of hand OA. It measures pain (5 questions), stiffness (1 question) and difficulties with daily activities (9 questions) through a visual analogue scale (0-100mm; 0 = lowest score; 100 = highest score). Lower AUSCAN scores represent a better outcome. Change (from baseline to month 24) in these scores was calculated.
Time Frame: Baseline and Month 24
Population: About 15% of the ITT population had hand OA at baseline and only these subjects were included in the X-ray assessments.The AUSCAN questionnaire was administered to all the patients at sites in Denmark, the Czech Republic, and Romania.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 585 | 584
Scores on a scale
  Total osteophytes: number analyzed (Participants) | 58 | 64
  Total osteophytes | 0.40 (0.784) | 0.40 (0.754)
  Total JSN: number analyzed (Participants) | 58 | 64
  Total JSN | 0.45 (1.063) | 0.62 (0.990)
  Total cyst/erosions: number analyzed (Participants) | 58 | 64
  Total cyst/erosions | 0.83 (1.204) | 0.82 (1.327)
  Total osteophytes, JSN and cyst/erosions: number analyzed (Participants) | 58 | 64
  Total osteophytes, JSN and cyst/erosions | 1.68 (2.682) | 1.84 (2.714)
  AUSCAN total score: number analyzed (Participants) | 297 | 330
  AUSCAN total score | -51.5 (265.13) | -38.1 (272.07)

6. Secondary Outcome: Nature and # of AEs Monitored Continuously During Study
Description: Adverse events were by system organ class of all patients.
Time Frame: From Baseline to Month 24
Population: ITT population. A patient with multiple occurrences of a TEAE under one treatment is counted only once in the AE category for that treatment.
Measure: Number; unit: Number of AEs by system organ class
Groups:
- Total: Total number of subjects between the two groups
Arm/Group | Active Arm | Placebo Arm | Total
Number analyzed (Participants) | 585 | 584 | 1169
Number of AEs by system organ class
  Any primary system organ class | 548 | 520 | 1068
  Blood and lymphatic system disorders | 18 | 16 | 34
  Cardiac disorders | 38 | 30 | 68
  Congenital, familial and genetic disorders | 1 | 0 | 1
  Ear and labyrinth disorders | 14 | 12 | 26
  Endocrine disorders | 9 | 9 | 18
  Eye disorders | 17 | 22 | 39
  Gastrointestinal disorders | 268 | 150 | 418
  General disorders and administration site condit. | 60 | 53 | 113
  Hepatobiliary disorders | 11 | 10 | 21
  Immune system disorders | 8 | 4 | 12
  Infections and infestations | 231 | 249 | 480
  Injury, poisoning and procedural complications | 87 | 95 | 182
  Investigations | 53 | 53 | 106
  Metabolism and nutrition disorders | 76 | 64 | 140
  Musculoskeletal and connective tissue disorders | 231 | 267 | 498
  Neoplasms benign, malignant and unspecified | 27 | 16 | 43
  Nervous system disorders | 96 | 87 | 183
  Psychiatric disorders | 28 | 27 | 55
  Renal and urinary disorders | 19 | 14 | 33
  Reproductive system and breast disorders | 18 | 20 | 38
  Respiratory, thoracic and mediastinal disorders | 48 | 49 | 97
  Skin and subcutaneous tissue disorders | 69 | 36 | 105
  Surgical and medical procedures | 27 | 30 | 57
  Vascular disorders | 160 | 92 | 252

7. Secondary Outcome: Disease Progression in the Knee Evaluated by MRI.
Description: Disease progression in the signal knee (cartilage volume and thickness) were evaluated by magnetic resonance imaging (MRI). MRIs were performed for patients from the sites in Ballerup, Denmark, the Czech Republic, and Romania using a quality controlled low-field 0.18T C-Span scanner from Esaote dedicated to the imaging of extremities. The same solenoid coil was used for all patients at a given site.
Time Frame: From Baseline to Month 24
Population: MRIs were performed for patients from the sites in Ballerup, Denmark, the Czech Republic, and Romania.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 268 | 261
percentage of change
  Total cartilage volume m12: number analyzed (Participants) | 194 | 216
  Total cartilage volume m12 | 2.90 (10.104) | 0.26 (9.283)
  Total cartilage volume m24: number analyzed (Participants) | 172 | 203
  Total cartilage volume m24 | 4.79 (10.352) | 1.94 (9.257)
  Total cartilage thickness m12: number analyzed (Participants) | 194 | 216
  Total cartilage thickness m12 | 1.9921 (7.05068) | 0.4343 (6.90177)
  Total cartilage thickness m24: number analyzed (Participants) | 172 | 203
  Total cartilage thickness m24 | 3.1777 (6.22356) | 2.2467 (7.09590)

ADVERSE EVENTS:
Time Frame: From baseline until 30 days following the end of study.
Description: The safety population is all patients randomized who received at least one dose of study medication. There were 7 patients in the randomized population who did not receive any study drug and where therefore excluded from the safety analysis.
Arm/Group | Active Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 100/585 | 88/584
Other Adverse Events (participants affected / at risk) | 548/585 | 520/584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Arm (N=585) | Placebo Arm (N=584)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 12
Bone graft (Surgical and medical procedures) | 4 | 7
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 5 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 3
Chest pain (General disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 3 | 0
Obesity (Metabolism and nutrition disorders) | 3 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Colonic polyp (Gastrointestinal disorders) | 2 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Knee arthroplasty (Surgical and medical procedures) | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Coronary artery dilatation (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Accidental death (General disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leimyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urethral prolapse (Renal and urinary disorders) | 0 | 1
Urinary retension (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peau d´orange (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Abscess drainage (Surgical and medical procedures) | 1 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1
Cardial pacemaker insertion (Surgical and medical procedures) | 0 | 1
Gastric bypass (Surgical and medical procedures) | 1 | 0
Lipoma excision (Surgical and medical procedures) | 0 | 1
Radical hysterectomy (Surgical and medical procedures) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Arm (N=585) | Placebo Arm (N=584)
Arthralgia (Musculoskeletal and connective tissue disorders) | 89 | 93
Hot flush (Vascular disorders) | 104 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 62 | 59
Nausea (Gastrointestinal disorders) | 82 | 18
Hypertension (Vascular disorders) | 46 | 52
Nasopharyngitis (Infections and infestations) | 43 | 55
Influenza (Infections and infestations) | 36 | 52
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 36 | 52
Dyspepsia (Gastrointestinal disorders) | 59 | 26
Diarrhoea (Gastrointestinal disorders) | 56 | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 | 30
Hypercholesterolemia (Metabolism and nutrition disorders) | 30 | 36
Headache (Nervous system disorders) | 35 | 28
Cystitis (Infections and infestations) | 35 | 17
Pneumonia (Infections and infestations) | 28 | 24
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 | 30
Procedural pain (Injury, poisoning and procedural complications) | 29 | 20
Abdominal pain upper (Gastrointestinal disorders) | 26 | 20
Dizziness (Nervous system disorders) | 18 | 25
Upper respiratory tract infection (Infections and infestations) | 18 | 19
Bronchitis (Infections and infestations) | 15 | 19
Sinusitis (Infections and infestations) | 17 | 15
Viral infections (Infections and infestations) | 10 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Tooth infection (Infections and infestations) | 19 | 10
Erythema (Skin and subcutaneous tissue disorders) | 25 | 3
Influenza like illness (General disorders) | 16 | 12
Contusion (Injury, poisoning and procedural complications) | 13 | 11
Fatigue (General disorders) | 10 | 14
Gastroenteritis (Infections and infestations) | 10 | 14
Oedema peripheral (General disorders) | 10 | 14
Abdominal pain (Gastrointestinal disorders) | 12 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 13 | 9
Depression (Psychiatric disorders) | 14 | 7
Constipation (Gastrointestinal disorders) | 13 | 7
Joint sprain (Injury, poisoning and procedural complications) | 8 | 12
Rash (Skin and subcutaneous tissue disorders) | 12 | 6
Vomiting (Gastrointestinal disorders) | 13 | 5
Abdominal discomfort (Gastrointestinal disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days